CLINICAL TRIAL: NCT04777513
Title: Evaluation of Diagnostic Accuracy, Safety, and Cost-Effectiveness of the Non-Invasive Cardiolens FFR-CT Pro Method to Measure the Fractional Flow Reserve in Diagnostics of Chronic Coronary Syndromes Versus the Standard Diagnostic Modalities. A Multicentre Post-marketing Trial of a Class 2a Medical Device, Cardiolens FFR-CT Pro - Software for Non-invasive Determination of Haemodynamic Parameters in Coronary Arteries.
Brief Title: Evaluation of Diagnostic Accuracy, Safety, and Cost-Effectiveness of the Non-Invasive Cardiolens FFR-CT Pro Method to Measure the Fractional Flow Reserve in Diagnostics of Chronic Coronary Syndromes Versus the Standard Diagnostic Modalities.
Status: Completed | Type: Observational
Sponsor: Hemolens Diagnostics Sp. z o.o. (Other)
Collaborators: GENELYTICA Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Other Study IDs: HEMOFLOW PMS_2020
Record Dates: First submitted 2021-02-08; First posted 2021-03-02 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stable Ischemic Heart Disease; Coronary Artery Disease
Keywords: Fractional Flow Reserve; Chronic Coronary Syndromes; Coronary Artery lesions; Vascular Diseases; Post-market surveillance; Invasive Coronary Angiography; Coronary Computed Tomography Angiography
MeSH Terms: conditions — Coronary Artery Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Standard of care: FFR, ICA, CCTA: Patients with medical history for ischaemic heart disease will take part in non-invasive determination of haemodynamic parameters in coronary arteries with Cardiolens FFR-CT Pro technology.
  Interventions: Procedure: CCTA (Coronary Computed Tomography Angiography); Procedure: ICA (Invasive Coronary Angiography); Procedure: FFR (Fractional Flow Reserve); Device: CNBP measurement; Device: Cardiolens FFR-CT Pro

INTERVENTIONS:
Procedure: CCTA (Coronary Computed Tomography Angiography) — Per the protocol, patients had a coronary computed tomography angiography within standard of care before the enrollment to the study.
Procedure: ICA (Invasive Coronary Angiography) — Per the protocol, patients will have an Invasive Coronary Angiography within standard of care.
Procedure: FFR (Fractional Flow Reserve) — Per the protocol, patients will have a Fractional Flow Reserve procedure within standard of care.
Device: CNBP measurement — Per the protocol, patients will have the measurement of the resting Continuous Non-Invasive Blood Pressure (CNBP). The signal is required for iSIL-FFR technology.
Device: Cardiolens FFR-CT Pro — Per the protocol, non-invasive FFR measurements will be perfomed via Cardiolens FFR-CT Pro technology for the enrolled patients.

SUMMARY:
A multicentre, post-marketing, observational trial in 450 patients, whose standard diagnostic workup for chronic coronary syndromes provided for Invasive Coronary Angiography (ICA). Medical records of a potential subject of the trial before their enrolment contain a good quality result of at least 128-slice CCTA performed up to 3 months before the elective ICA. CCTA should find at least one ≥50% stenosis in at least one big coronary artery of ≥ 2 mm diameter. At one hour before ICA in the latest the patient should have a resting Continuous Non-Invasive Blood Pressure (CNBP) taken with a certified device delivered by LifeFlow. The last criterion before including a patient in the final analysis is at least one significant (≥50%) stenosis in one or two coronary arteries of ≥ 2 mm diameter visually confirmed by ICA with a FFR measurement taken in these arteries.

The data collection period will cover time from admission for the elective ICA to discharge from the hospital (evaluation of possible adverse events related to invasive procedures).

After initial qualification of available data by the attending physician, selected patients will be asked for a consent to participation in the trial no later than upon admission for the elective ICA and before CNBP measurement.

DETAILED DESCRIPTION:
Stage 1

After a patient declares their consent, a doctor or another member of the study team trained by the sponsor will perform procedures in the following order:

* Define the unique patient ID to be recorded in the CRF with the patient's demographic data
* Assess the quality of CCTA imaging data (DICOM) according to guidelines agreed upon with the sponsor and record the number and location of the significant (≥50%) stenosis sites in the CRF based on CCTA
* No later than one hour before ICA starts, perform a physical examination consisting in instantaneous peripheral blood pressure (systolic and diastolic) resting measurement performed with a standard sphygmomanometer and Continuous Non-Invasive Blood Pressure measurement (1-3 min).

Stage 2

After the procedures mentioned above are performed, the patient will undergo elective ICA with the outcomes, i.e.:

* video material showing the location of the wire during the FFR measurement,
* digital pressure signals exported from the FFR measuring device used to determine the value of the invasive FFR,
* values of FFR measurements obtained during ICA will be entered after being anonymised in a dedicated HEMOFLOW PMS_2020 reference database.

Stage 3

Within 48 hours of ICA completion a doctor or another member of the study team trained by the sponsor:

* will enter the following data in the Cardiolens FFR-CT Pro system:

  1. Patient's data, i.e. patient's ID, gender, height, body mass, exercise tolerability, information on used medications and smoking cigarettes. Optionally, i.e. if upon admission for ICA a blood test was performed as a part of the standard diagnostic workup - haematocrit levels and total protein concentration
  2. Files containing CCTA imaging data in the DICOM format.
  3. Values of instantaneous peripheral blood pressure (systolic and diastolic) resting measurement performed with a standard sphygmomanometer as well as the digital signal obtained during the CNBP measurement (1-3 min)
* Based on the CCTA description or meta data contained in the imaging data the doctor or another member of the study team will record the following information in the CRF:

  1. Radiation dose during CCTA
  2. Contrast medium dose during CCTA
* Will enter the following information in the CRF:

  1. Radiation dose during the diagnostic part of ICA
  2. Contrast medium dose during the diagnostic part of ICA
  3. Number and type of adverse events
  4. Duration of the diagnostic workup.

Stage 4

Within 7 days of entering all the stage 3 data the investigator (a cardiologist) trained by the sponsor will measure the value of the virtual FFR with the Cardiolens FFR-CT Pro system at locations corresponding to ICA FFR measurements (based on video recording entered in the database during stage 2)

Based on results obtained from the Cardiolens FFR-CT Pro system vs reference data an analysis will be performed on meeting the primary and secondary end points of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Declaration of informed consent to sharing medical records gathered during the standard diagnostic workup
3. History of chronic coronary syndromes (CCS)
4. Diagnostic CCTA (good quality test allowing investigation of the entire coronary artery tree), showing at least one site with stenosis ≥50% of the lumen in a large coronary artery of ≥ 2 mm diameter, with no prior revascularisation
5. Standard treatment of chronic coronary syndromes with no dosage modification required within at least 4 weeks before the enrolment
6. Patients with a prior acute coronary syndrome (ACS) or revascularisation would be found eligible under the following conditions:

   * Over 30 days from the acute coronary syndrome occurrence
   * FFR assessment during ICA may only cover the vessels that were not revascularized (both PCI and CABG) and were not the reason of ACS
   * No closed coronary arteries

Exclusion Criteria:

1. CCTA-confirmed myocardial bridges causing >50% stenosis of the epicardial vascular lumen
2. Coronary obstruction confirmed by CCTA or invasive coronarography
3. History of ACS with coronary angioplasty or Coronary Artery Bypass Grafting (CABG) performed unless point 6 conditions are met
4. Significant haemodynamic abnormalities of the valve or history of surgical correction of the defect or CABG
5. Second-degree or third-degree atrioventricular block, sinus node dysfunction, QTc > 450 ms or prolonged QTc
6. LVEF ≤ 35% found in an echocardiogram performed within the last 6 months
7. BMI ≥ 35
8. Clinically apparent infection
9. Thrombocytopenia below 100.000/mm3
10. Active neoplastic disease (apart from basal cell carcinoma and carcinoma in situ) and other conditions, which, in the investigator's opinion significantly affect their life expectancy
11. Other significant conditions, infections, addictions and psychological or social factors, which, in the doctor's opinion, may affect patient's ability to participate in the trial or significantly affect their safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the trial are patients, who will undergo standard diagnostic workup for chronic coronary syndromes (including standard procedures according to valid 2019 ESC guidelines, i.e. medical history for ischaemic heart disease, CCTA, and ICA with FFR as indicated) as a part of health care services.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The evaluation of the increased diagnostic accuracy of the non-invasive Cardiolens FFR-CT Pro technology | Up to 18 months
  Evaluation of the increased diagnostic accuracy (area under ROC curve, AUC) in detection of haemodynamically significant stenoses in coronary arteries with a non-invasive Cardiolens FFR-CT Pro technology compared to CCTA in reference to the invasive fractional flow reserve (FFR) testing at the arterial level.

SECONDARY OUTCOMES:
The evaluation of diagnostic accuracy of the non-invasive Cardiolens FFR-CT Pro technology | Up to 18 months
  Evaluation of diagnostic accuracy of Cardiolens FFR-CT Pro in detection of haemodynamically significant stenoses in coronary arteries (FFR value ≤0.80) compared to CCTA (stenosis ≥ 50%), in reference to the invasive FFR testing at the patient and arterial level, based on parameters like sensitivity, specificity, positive/negative predictive value, accuracy at the patient and arterial level.
The evaluation of safety of the non-invasive Cardiolens FFR-CT Pro technology | Up to 5 days. The date from admission for the scheduled ICA to discharge from the hospital.
  Evaluation of safety of the non-invasive Cardiolens FFR-CT Pro technology (the result of the non-invasive test completes the diagnostic workup for coronary disease) compared to the standard diagnostics in chronic coronary syndromes based on the following parameters:
  1. Radiation dose during the diagnostic workup
  2. Contrast medium dose in the diagnostic workup
  3. Adverse events during the diagnostic workup
  4. Duration of the diagnostic workup
The evaluation of the costs of Cardiolens FFR-CT Pro technology | Up to 5 days. The date from admission for the scheduled ICA to discharge from the hospital.
  3) Evaluation of the costs of Cardiolens FFR-CT Pro in diagnostics of chronic coronary syndromes compared to the standard diagnostic workup (the sum of the costs for individual diagnostic modalities according to the National Health Fund reimbursement prices as well as Procedural Reimbursement Payment Guide)

CONTACTS AND LOCATIONS:
Overall Officials: Cezary Kępka, MD, PhD, Principal Investigator — The National Institute of Cardiology
Locations (11):
- Poland (11):
  - American Heart of Poland, Centrum Kardiologii i Kardiochirurgii w Bielsku-Białej, Bielsko-Biala
  - The University Clinical Centre, Gdansk
  - The Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University, Katowice
  - Oddział Kliniczny Kardiologii oraz Interwencji Sercowo-Naczyniowych Szpital Uniwersytecki w Krakowie, Krakow
  - The John Paul II Specialist Hospital in Cracovia, Krakow
  - "Miedziowe Centrum Zdrowia" S.A., Lubin
  - American Heart of Poland, Centrum Sercowo - Naczyniowe w Ustroniu, Ustroń
  - The Cardinal Stefan Wyszyński National Institute of Cardiology, Warsaw
  - The 4th Military Teaching Hospital, Wroclaw
  - The Jan Mikulicz-Radecki University Teaching Hospital, Wroclaw
  - The T. Marciniak Lower Silesian Specialist Hospital - Center of Emergency Medicine, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213
- [Background] Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Uva MS, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A; Grupa Robocza Europejskiego Towarzystwa Kardiologicznego (ESC); Europejskie Stowarzyszenie Chirurgii Serca i Klatki Piersiowej (EACTS) do spraw rewaskularyzacji miesnia sercowego; European Association for Percutaneous Cardiovascular Interventions (EAPCI). [2014 ESC/EACTS Guidelines on myocardial revascularization]. Kardiol Pol. 2014;72(12):1253-379. doi: 10.5603/KP.2014.0224. No abstract available. Polish. PMID 25524605
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Lindstaedt M, Fritz MK, Yazar A, Perrey C, Germing A, Grewe PH, Laczkovics AM, Mugge A, Bojara W. Optimizing revascularization strategies in patients with multivessel coronary disease: impact of intracoronary pressure measurements. J Thorac Cardiovasc Surg. 2005 Apr;129(4):897-903. doi: 10.1016/j.jtcvs.2004.08.036. PMID 15821661
- [Background] Reczuch K, Jankowska E, Telichowski A, Porada A, Banasiak W, Ponikowski P. Measurement of fractional flow reserve in patients with multi-vessel coronary artery disease and borderline lesions prevents unnecessary revascularisation procedures. Kardiol Pol. 2004 Apr;60(4):311-19; discussion 320-1. English, Polish. PMID 15226780
- [Background] Toth G, De Bruyne B, Casselman F, De Vroey F, Pyxaras S, Di Serafino L, Van Praet F, Van Mieghem C, Stockman B, Wijns W, Degrieck I, Barbato E. Fractional flow reserve-guided versus angiography-guided coronary artery bypass graft surgery. Circulation. 2013 Sep 24;128(13):1405-11. doi: 10.1161/CIRCULATIONAHA.113.002740. Epub 2013 Aug 28. PMID 23985788
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] De Bruyne B, Pijls NH, Barbato E, Bartunek J, Bech JW, Wijns W, Heyndrickx GR. Intracoronary and intravenous adenosine 5'-triphosphate, adenosine, papaverine, and contrast medium to assess fractional flow reserve in humans. Circulation. 2003 Apr 15;107(14):1877-83. doi: 10.1161/01.CIR.0000061950.24940.88. Epub 2003 Mar 31. PMID 12668522
- [Background] Wongpraparut N, Yalamanchili V, Pasnoori V, Satran A, Chandra M, Masden R, Leesar MA. Thirty-month outcome after fractional flow reserve-guided versus conventional multivessel percutaneous coronary intervention. Am J Cardiol. 2005 Oct 1;96(7):877-84. doi: 10.1016/j.amjcard.2005.05.040. PMID 16188509
- [Background] Leone AM, Martin-Reyes R, Baptista SB, Amabile N, Raposo L, Franco Pelaez JA, Trani C, Cialdella P, Basile E, Zimbardo G, Burzotta F, Porto I, Aurigemma C, Rebuzzi AG, Faustino M, Niccoli G, Abreu PF, Slama MS, Spagnoli V, Telleria Arrieta M, Amat Santos IJ, de la Torre Hernandez JM, Lopez Palop R, Crea F. The Multi-center Evaluation of the Accuracy of the Contrast MEdium INduced Pd/Pa RaTiO in Predicting FFR (MEMENTO-FFR) Study. EuroIntervention. 2016 Aug 20;12(6):708-15. doi: 10.4244/EIJV12I6A115. PMID 27542782
- [Background] Wu W, Pan DR, Foin N, Pang S, Ye P, Holm N, Ren XM, Luo J, Nanjundappa A, Chen SL. Noninvasive fractional flow reserve derived from coronary computed tomography angiography for identification of ischemic lesions: a systematic review and meta-analysis. Sci Rep. 2016 Jul 5;6:29409. doi: 10.1038/srep29409. PMID 27377422
- [Background] Nakazato R, Park HB, Berman DS, Gransar H, Koo BK, Erglis A, Lin FY, Dunning AM, Budoff MJ, Malpeso J, Leipsic J, Min JK. Noninvasive fractional flow reserve derived from computed tomography angiography for coronary lesions of intermediate stenosis severity: results from the DeFACTO study. Circ Cardiovasc Imaging. 2013 Nov;6(6):881-9. doi: 10.1161/CIRCIMAGING.113.000297. Epub 2013 Sep 30. PMID 24081777
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Morris PD, van de Vosse FN, Lawford PV, Hose DR, Gunn JP. "Virtual" (Computed) Fractional Flow Reserve: Current Challenges and Limitations. JACC Cardiovasc Interv. 2015 Jul;8(8):1009-1017. doi: 10.1016/j.jcin.2015.04.006. Epub 2015 Jun 24. PMID 26117471
- [Background] Kruk M, Wardziak L, Demkow M, Pleban W, Pregowski J, Dzielinska Z, Witulski M, Witkowski A, Ruzyllo W, Kepka C. Workstation-Based Calculation of CTA-Based FFR for Intermediate Stenosis. JACC Cardiovasc Imaging. 2016 Jun;9(6):690-9. doi: 10.1016/j.jcmg.2015.09.019. Epub 2016 Feb 17. PMID 26897667
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- See also: WHO Fact sheet N°317 September 2012 — http://www.who.int/mediacentre/factsheets/fs317/en/
- See also: WHO Fact sheet N°310 Updated June 2011 — http://who.int/mediacentre/factsheets/fs310/en/
- See also: Related Info — http://ec.europa.eu/growth/sectors/medical-devices/contacts/
- See also: Related Info — http://www.urpl.gov.pl/pl/wyroby-medyczne/informacje-dotyczące-bezpieczeństwa/formularze